CLINICAL TRIAL: NCT01148394
Title: Impact of the Introduction of a Multimodal Rehabilitation Programme for Colorectal Patients. A Prospective Randomized Trial.
Brief Title: Enhanced Recovery After Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Stephanie Garcia Botello, Hospital Clinico Universitario, Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT-1
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Fast Track; Enhanced Recovery
Keywords: Colorectal surgery; multimodal rehabilitation; fast track; early feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional (No Intervention): Involves traditional management of patients with preoperative mechanical bowel preparation, no preoperative education, nasogastric tube, delayed feeding and mobilisation, use of drains
  Interventions: Other: Multimodal rehabilitation
- Multimodal rehabilitation (Active Comparator): Involves preoperative patient education, no preoperative mechanical bowel preparation, no nasogastric tube, early oral feeding and mobilisation, physiotherapy
  Interventions: Other: Multimodal rehabilitation

INTERVENTIONS:
Other: Multimodal rehabilitation

SUMMARY:
Introduction: Multimodal rehabilitation (MMR), combines various elements in the management of the surgical patient which lead to a decrease in surgical stress and a more comfortable and faster postoperative recovery.

Objective: To assess the introduction of MMR in a specialized Colorectal Unit and compare the results with the traditional model assessing its´ efficacy as to recovery, and reduction of hospital stay and costs.

DETAILED DESCRIPTION:
Materials y Methods: A prospective randomized trial was conducted which analyzed 119 patients who underwent elective colorectal surgery between 2009 and 2010. 58 patients were assigned to the traditional group and 61 patients to the MMR group. MMR included preoperative education, early feeding and mobilisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective colorectal surgery between 2009 and 2010.
* Signed informed consent
* Live in Valencia metropolitan area

Exclusion Criteria:

* Emergency surgery
* No colonic resection
* Unable to continue follow-up
* Dependent on others for daily activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Postoperative stay | 18 months

SECONDARY OUTCOMES:
Postoperative complications | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Garcia Botello, MBChB, Principal Investigator — Hospital Clinico Universitario Valencia; Eduardo Garcia-Granero, MD, Study Chair — Hospital Clinico Universitario, Valencia

REFERENCES:
- [Derived] Garcia-Botello S, Canovas de Lucas R, Tornero C, Escamilla B, Espi-Macias A, Esclapez-Valero P, Flor-Lorente B, Garcia-Granero E. [Implementation of a perioperative multimodal rehabilitation protocol in elective colorectal surgery. A prospective randomised controlled study]. Cir Esp. 2011 Mar;89(3):159-66. doi: 10.1016/j.ciresp.2010.12.004. Epub 2011 Feb 22. Spanish. PMID 21345423